CLINICAL TRIAL: NCT04259684
Title: Efficacy of Nitric Oxide Administration During Cardiopulmonary Bypass in Neonates at Reducing the Risk of Acute Kidney Injury: a Preliminary Double-blind Randomized Controlled Trial
Brief Title: Nitric Oxide During Cardiopulmonary Bypass in Neonates to Reduce Risk of Acute Kidney Injury
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: revised and combined with another protocol
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIN001-gNO to prevent AKI
Record Dates: First submitted 2019-03-19; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury; Congenital Heart Disease
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Each of the 40 participants will be stratified based on type of lesion (single ventricle vs. biventricular lesions) and block randomized into 1 of 2 study arms: treatment arm (receiving intraoperative administration of 20 ppm of gNO to the oxygenator of the CPB circuit) and control arm (standard CPB conduct).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- gNO Group (Experimental): Participants in the treatment group will receive gNO added to the oxygenator gas flow at 20 ppm throughout the duration of cardiopulmonary bypass.
  Interventions: Drug: gases Nitric Oxide (gNO)
- Control Group (No Intervention): Participants in the control group will receive standard conduction of cardiopulmonary bypass.

INTERVENTIONS:
Drug: gases Nitric Oxide (gNO) — Participants in the intervention group will receive gNO blended into the fresh gas flow of the cardiopulmonary bypass (CPB) oxygenator and maintained at 20 ppm via an Ikaria INO Max DSIR (Mallinckrodt Pharmaceuticals, St. Louis, Missouri, USA), with continuous sampling of NO and NO2 concentration from a port adjacent to the oxygenator. The gNO delivery will be initiated when the patient is on CPB and stopped once the patient comes off CPB.
  Arms: gNO Group

SUMMARY:
Acute kidney injury following cardiac surgery for congenital heart defects in children is a major cause of both short- and long-term morbidity and mortality, affecting up to 60% of high risk patients. Despite effort, to date, no successful therapeutic agent has gained widespread success in preventing this postoperative decline in renal function. Based on preliminary data available in the literature, we hypothesize that nitric oxide (gNO), administered during cardiopulmonary bypass (CPB), may reduce the risk of acute kidney injury (AKI) via mechanisms of reduced inflammation and vasodilation. In this pilot study, 40 neonates undergoing cardiac surgery will be randomized to receive intraoperative administration of 20 ppm of nitric oxide to the oxygenator of the cardiopulmonary bypass circuit or standard CPB with no additional gas.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (≤31 days) undergoing cardiac surgery with cardiopulmonary bypass for congenital heart disease

Exclusion Criteria:

* 1. Failure to obtain informed consent from parent/guardian,
* Clinical signs of preoperative persistent elevated pulmonary vascular resistance,
* Emergency surgery,
* Episode of cardiac arrest within 1 week before surgery,
* Recent treatment with steroids and/or a condition that may require treatment with steroids (excluding steroid administration specifically for CPB),
* Use of inhaled NO (iNO) immediately prior to surgery,
* Structural renal abnormalities by ultrasound,
* Preoperative AKI,
* Use of other investigational drugs,
* Weight less than <2.2 kg,
* Gestational age <36 weeks,
* Major extracardiac congenital anomalies.

Max Age: 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | up to 72 hours postoperative
  Occurrence of acute kidney defined by the Kidney Disease Improving Global Outcomes (KDIGO) diagnostic classification (employing both serum creatinine and urine output criteria).
Glomerular Filtration Rate | up to 72 hours postoperative
  Postoperative glomerular filtration rate (GFR) measured using serum cystatin C.

SECONDARY OUTCOMES:
Structural Kidney Injury | up to 72 hours postoperative
  Assessed by measurement of urine biomarkers: neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecule-1 (KIM-1), interleukin-18 (IL-18) liver-type fatty acid-binding protein (L-FABP), and urinary nitrate.
Low cardiac output syndrome (LCOS) | up to 48 hours postoperative
  Occurence of low cardiac output syndrome (LCOS) defined as any of the following at any time during the first 48 hours postoperative:
  1. Lactate >6mmol/l and central venous saturation (ScvO2) <60% (or SaO2-ScvO2 difference greater than 35% in a single ventricle),
  2. Vasoactive inotropic score (VIS)24 ≥ 10,
  3. Extracorporeal Membrane Oxygenation (ECMO).
Duration of mechanical ventilation | up to 2 weeks from admission to CICU to extubation
  hours/days
Length of cardiac intensive care unit (CICU) stay | up to 2 weeksfrom admission to CICU to discharge from CICU
  days
Length of hospital stay | up to 30 days from hospital admission to discharge
  days
Inotrope free days | up to 30 days after surgery to CICU discharge
  days
ECMO free days | up to 2 weeks after surgery to CICU discharge
  Extracorporeal Membrane Oxygenation free days
Closed sternum days | up to 2 weeks from postoperative CICU admission to discharge
  days
Time to negative fluid balance | up to 2 weeks from CICU admission to outcome reached
  hours/days
Urine Output | up to two weeks from CICU admission to discharge
  ml
Use of peritoneal dialysis | up to two weeks from CICU admission to discharge
  yes/no
Cardiac arrest | up to two weeks from CICU admission to discharge
  yes/no
Use of postoperative inhaled Nitric Oxide (iNO) | up to two weeks from CICU admission to discharge
  yes/no, indication, dose

IPD SHARING:
Plan to Share IPD: No